CLINICAL TRIAL: NCT02295592
Title: TSTstarr + for Treatment of Severe Prolapsed Hemorrhoids --- a Multi-center Randomized Controlled Clinical Trail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Suzhou Touchstone International Medical Science Co.,Ltd. (Unknown); Chengdu Anorectal Hospital (Unknown); Wuhan University (Other); Fujian Provincial Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Nanhai Hospital of Traditional Chinese Medicine (Other); Changshu Hospital of Traditional Chinese Medicine (Other); Xuzhou Central Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Shenyang Anorectal Hospital (Other); Wulumuqi General Hospital of Lanzhou Military Command (Other); The First Affiliated Hospital of Guangxi traditional Chinese Medicine University (Unknown); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014ZSLYEC-021
Record Dates: First submitted 2014-11-05; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-10

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids; The recurrence rate; PPH; TSTstarr+
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A( TSTstarr+ group) (Experimental): TSTstarr+ is a kind of modified STARR（stapled transanal rectal resection ） operation, compared to the traditional STARR operation, it does not need two staplers but with a larger diameter stapler, " +" means better . Patients in group A with severe prolapsed hemorrhoids will undergo TSTstarr+ operation .
  Interventions: Procedure: TSTstarr+
- group B ( PPH group) (Active Comparator): PPH is short fo procedure for prolapsed hemorrhoids .Patients in group B with severe prolapsed hemorrhoids will undergo PPH operation.
  Interventions: Procedure: PPH

INTERVENTIONS:
Procedure: TSTstarr+ — TSTstarr+ : a kind of modified STARR（stapled transanal rectal resection ） operation, compared to the traditional STARR operation, it does not need two staplers but with a larger diameter stapler, " +" means better . Patients in group A with severe prolapsed hemorrhoids will undergo TSTstarr+ operation .
  Arms: group A( TSTstarr+ group)
Procedure: PPH — PPH is short fo procedure for prolapsed hemorrhoids .Patients in group B with severe prolapsed hemorrhoids will undergo PPH operation.
  Arms: group B ( PPH group)

SUMMARY:
TSTstarr+ in the treatment of severe hemorrhoids prolapse--A multi center randomized controlled clinical trial.The aim of this stuy is to compare the first year hemorrhoids recurrence rate of TSTstarr+ and PPH in the treatment of severe hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

* severe prolapsed hemorrhoids
* no significant anal-malformation before operation
* having signed the informed consent.

Exclusion Criteria:

* needing emergency operation or having previous history of hemorrhoids operation
* with other anal diseases at the same time such as : anal fissure, anal fistula and perianal abscess and so on
* diagnosed with inflammatory bowel disease or proctitis
* diagnosed with colorectal cancer
* associated with cardiovascular and cerebrovascular diseases and other diseases so that can not tolerate surgery or increase the risk of surgery
* with chronic or acute renal insufficiency patients
* coagulation abnormalities or with anticoagulation treatment at present
* diagnosed with diabetes with poor glycemic control
* in women with pregnant or menstruation
* The intellectual disabilities or mental disorder
* had participated in other clinical trial before we selected 4 weeks
* other severe complications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-04 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
the recurrence rate of the severe prolapsed Hemorrhoids after surgery | 2 years
  780 patients will be enrolled in one year.All patients will be followed up for one year, and then calculate 1 year recurrence rate between TSTstarr+ group and PPH group

SECONDARY OUTCOMES:
Operation time | 1 year
Intraoperative hemorrhage | 1 year
The weight of specimens | 1year
The volume of specimens | 1year
The number of patients with anal pain after surgery | 2 years
The number of patients with fecal urgency after surgery | 2 years
The number of patients with stricture of anus after surgery | 2 years
The number of patients with hemorrhage after surgery | 2 years
The number of patients with retention of urine in the early time after surgery | 2 years
The number of patients with edema of the anal margin in the early time after surgery | 2 years
The time of returning to normal | 2 years
The total cost of hospitalization | 2 years